CLINICAL TRIAL: NCT02484729
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Access the Safety, Tolerability and Pharmacokinetics of AZD9977 Following Single Ascending Dose Administration to Healthy Male Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD9977 After Single Ascending Doses to Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D6400C00001; 2015-000877-11 (EudraCT Number)
Record Dates: First submitted 2015-06-18; First posted 2015-06-30 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Safety; Tolerability; Pharmacokinetics; Healthy Subjects
Keywords: AZD9977; Safety; Tolerability; Pharmacokinetics; First-in-human; Single Ascending Dose; Regional absorption; Healthy male subjects
MeSH Terms: interventions — AZD9977; Suspensions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD9977 oral suspension, single doses (Experimental): In Part A up to 10 cohorts with single ascending doses with AZD9977 as oral suspension. In Part B AZD9977 as oral suspension in IntelliCap® capsule
  Interventions: Drug: AZD9977, oral suspension
- Placebo, oral suspension, single doses (Placebo Comparator): In Part A up to 10 cohorts with single doses with matching placebo to AZD9977
  Interventions: Drug: Placebo, oral suspension
- AZD9977, oral solution, single dose (Experimental): In Part B, of oral solution of AZD9977 will be used as reference
  Interventions: Drug: AZD9977, oral solution

INTERVENTIONS:
Drug: AZD9977, oral suspension — Single ascending doses of AZD9977 oral suspension (Part A) Single dose of AZD9977 oral suspension in IntelliCap® capsule in regional absorption part (Part B)
  Arms: AZD9977 oral suspension, single doses
Drug: Placebo, oral suspension — Matching placebo
  Arms: Placebo, oral suspension, single doses
Drug: AZD9977, oral solution — AZD9977, single dose of oral solution in Part B as reference
  Arms: AZD9977, oral solution, single dose

SUMMARY:
This study will be a randomized, single-blind, placebo-controlled first-in-human study in healthy male subjects to assess the safety, tolerability and pharmacokinetics of single ascending doses of AZD9977. In Part B of this study the regional absorption of AZD9977 along the gastro-intestinal tract will be investigated using the IntelliCap® system in a non-randomized, open-label, fixed-sequence design. The study will be performed at a single study centre.

DETAILED DESCRIPTION:
This study will be a randomized, single-blind, placebo-controlled first-in-human study in healthy male subjects to assess the safety, tolerability and pharmacokinetics of single ascending doses of AZD9977. In Part B of this study the regional absorption of AZD9977 along the gastro-intestinal tract will be investigated using the IntelliCap® system in a non-randomized, open-label, fixed-sequence design with oral solution as reference. The study will be performed at a single study centre.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 18 to 50 years with suitable veins for cannulation or repeated venipuncture.
3. Male subjects have to comply with the restrictions for sexual activity provided to them.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Optional: Provision of signed and dated written informed consent for genetic research.

   If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.
6. Able to understand, read and speak the English language.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study, or influences the results or the potential subject's ability to participate in the study.
2. History or presence of GI, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of dosing in Part A or the first dose of AZD9977 in Part B.
4. Any clinically significant abnormalities in hematology, clinical chemistry or urinalysis results, as judged by the investigator.
5. Any positive result at screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody, and human immunodeficiency virus (HIV) antibodies.
6. Abnormal findings in vital signs, after 10 minutes resting in the supine position, defined as any of the following:

   * Systolic blood pressure (SBP) < 90 mmHg or ≥ 140 mmHg
   * Diastolic blood pressure (DBP) < 50 mmHg or ≥ 90 mmHg
   * Pulse < 45 or > 90 bpm
7. Any clinically important abnormalities in rhythm, conduction or morphology of the electrocardiogram (ECG) at screening or pre-dose, as considered by the investigator.
8. Prolonged QTcF > 450 ms or family history of long QT syndrome.
9. PR (PQ) interval shortening < 120 ms. PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation.
10. PR (PQ) interval prolongation > 240ms; intermittent second or third degree atrioventricular (AV) block, or AV dissociation.

    Wenckebach block while asleep is not exclusive.
11. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms.

    QRS > 110 ms but < 115 ms are acceptable if there is no evidence of ventricular hypertrophy or pre-excitation.
12. Serum potassium higher than 5.0 mmol/L at screening or admission to the study center (Day -1).
13. Known or suspected history of drug abuse as judged by the investigator.
14. Current smokers or those who have smoked or used nicotine products within the previous 3 months.
15. History of alcohol abuse or excessive intake of alcohol as judged by the investigator.
16. Positive screen for drugs of abuse, alcohol or cotinine at screening or admission to the study center.
17. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977.
18. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea and chocolate) as judged by the investigator.
19. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to dosing in Part A or the first dose of AZD9977 in Part B.
20. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during 2 weeks prior to dosing in Part A or the first dose of AZD9977 in Part B, or longer if the medication has a long half-life.
21. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.
22. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of dosing in Part A or the first dose of AZD9977 in Part B in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest.

    Note: Subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
23. Involvement of any AstraZeneca or study site employee or their close relatives.
24. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
25. Subjects who are vegans or have medical dietary restrictions (vegetarians may be included in the study).
26. Subjects who cannot communicate reliably with the investigator.
27. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

    In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
28. Previous bone marrow transplant.
29. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

    Criteria applicable to Part B only:
30. Subjects with pacemakers or other implanted electro-medical devices.
31. Subjects with swallowing disorders.
32. Subjects with pre-planned MRI examination.
33. Subjects not willing to have an abdominal X-ray performed if the IntelliCap® capsule has not been retrieved within one week after ingestion.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, Dr., Principal Investigator — PAREXEL Early Phase Clinical Unit London, Level 7, Northwick Park Hospital, Watford Road, Harrow, Middlesex HA1 3UJ, United Kingdom
Locations (1):
- Research Site, Harrow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL International, Early Phase Clinical Unit London, United Kingdom.
Pre-assignment Details: In this study, 196 subjects were screened out of which 70 subjects were randomized. The study was conducted in two parts (Parts A and B). Part A-eight cohorts of 8 subjects, randomized in 6:2 (AZD9977: placebo) and Part B -1 cohort of 8 subjects who received a single dose of AZD9977, on 2 occasions separated by washout period of 7 days.
Groups:
- Part A- Placebo: Subjects received matching placebo under fasted conditions
- Part A - 5 mg AZD9977: Subjects received 5 mg AZD9977, oral suspension under fasted conditions
- Part A - 25 mg AZD9977: Subjects received 25 mg AZD9977, oral suspension under fasted conditions
- Part A - 100 mg AZD9977: Subjects received 100 mg AZD9977, oral suspension under fasted conditions
- Part A - 200 mg AZD9977: Subjects received 200 mg AZD9977, oral suspension under fasted conditions
- Part A - 400 mg AZD9977: Subjects received 400 mg AZD9977, oral suspension under fasted conditions
- Part A - 800 mg AZD9977: Subjects received 800 mg AZD9977, oral suspension under fasted conditions
- Part A - 800 mg AZD9977 (Split Doses): Subjects received 800 mg AZD9977 (split doses), oral suspension under fasted conditions
- Part A - 1200 mg AZD9977 (Split Doses): Subjects received 1200 mg AZD9977 (split doses), oral suspension under fasted conditions
- Part B: Subjects received a single dose of AZD9977, under fasted conditions, on two occasions (40 mg AZD9977, IntelliCap device and 40 mg AZD9977, oral solution) separated by a washout period of at least 7 days
Period: Overall Study
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Started | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
Completed | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Failure of IntelliCap Error | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30 (6) | 32 (11) | 30 (9) | 36 (10) | 32 (10) | 33 (9) | 30 (6) | 32 (8) | 38 (11) | 35 (9) | 33 (9)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8 | 70

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of AZD9977 by Assessing the Percentage of Participants With Adverse Events
Description: To assess the safety and tolerability of single ascending doses of AZD9977
Time Frame: For up to 45 days, i.e. from Screening to Follow-up
Population: All subjects who received at least one dose of IMP and for whom any safety post-dose data were available were included in the safety analysis for the study.
Measure: Number; unit: percentage of participants
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
percentage of participants | 43.8 | 16.7 | 33.3 | 33.3 | 20.0 | 33.3 | 0 | 33.3 | 16.7 | 37.5

2. Primary Outcome: Safety and Tolerability of AZD9977 by Assessing Number of Participants With Clinically Significant Pulse Rate
Description: To assess the safety and tolerability of single ascending doses of AZD9977
Time Frame: For up to 45 days, i.e. from Screening to Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
Number of Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Safety and Tolerability of AZD9977 by Assessing Number of Participants With Clinically Significant Trends in 12-lead Electrocardiograms
Description: To assess the safety and tolerability of single ascending doses of AZD9977
Time Frame: For up to 45 days, i.e. from Screening to Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
Number of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Safety and Tolerability of AZD9977 by Number of Participants With Clinically Significant Trends in Cardiac Telemetry
Description: To assess the safety and tolerability of single ascending doses of AZD9977
Time Frame: For up to 4 days, i.e. on the day before each dosing and for 24 hours after each dosing
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
Number of Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Safety and Tolerability of AZD9977 by Assessing the Number of Subjects With Adverse Events
Description: To assess the safety and tolerability of single ascending doses of AZD9977
Time Frame: For up to 45 days, i.e. from Screening to Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
Number of Participants | 7 | 1 | 2 | 2 | 1 | 2 | 0 | 2 | 1 | 3

6. Primary Outcome: Safety and Tolerability of AZD9977 by Assessing Number of Participants With Clinically Significant Changes in Blood Pressure
Description: To assess the safety and tolerability of single ascending doses of AZD9977
Time Frame: For up to 45 days, i.e. from Screening to Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
Number of Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Safety and Tolerability of AZD9977 by Assessing Number of Participants With Clinically Significant Changes in Hematology
Description: To assess the safety and tolerability of single ascending doses of AZD9977
Time Frame: For up to 45 days, i.e. from Screening to Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
Number of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Safety and Tolerability of AZD9977 by Assessing Number of Participants With Clinically Significant Changes in Clinical Chemistry
Description: To assess the safety and tolerability of single ascending doses of AZD9977
Time Frame: For up to 45 days, i.e. from Screening to Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
Number of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Safety and Tolerability of AZD9977 by Assessing Number of Participants With Clinically Significant Changes in Urinalysis
Description: To assess the safety and tolerability of single ascending doses of AZD9977
Time Frame: For up to 45 days, i.e. from Screening to Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 8
Number of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Zero Extrapolated to Infinity.
Description: To assess plasma pharmacokinetic parameters following single ascending doses of AZD977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: The PK analysis set for Part A consisted of all subjects in the safety analysis set who received one dose of AZD9977 and had evaluable PK data. The PK analysis set for Part B consisted of all subjects in the safety analysis set who received at least one dose of AZD9977 and had evaluable PK data in at least one period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.nmol/L
Groups:
- Intellicap Device (Part B); Oral Suspension (Part B): Subjects received a single dose of AZD9977, under fasted conditions, on two occasions (40 mg AZD9977, IntelliCap device and 40 mg AZD9977, oral solution) separated by a washout period of at least 7 days
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Intellicap Device (Part B) | Oral Suspension (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 2 | 5 | 4 | 4 | 7
h.nmol/L | 514.4 (13.4) | 2473 (24.5) | 9576 (51.9) | 23810 (33.7) | 36210 (28.5) | 38060 (37.2) | 98910 (29.7) | 105700 (30.5) | 2256 (32.6) | 3294 (32.9)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Analyte concentrationAUC(0-t)
Description: To assess plasma pharmacokinetic parameters following single ascending doses of AZD977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.nmol/L
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Intellicap Device (Part B) | Oral Suspension (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 7 | 6
h.nmol/L | 482.7 (14.9) | 2429 (24.7) | 9419 (52.2) | 23470 (34.2) | 35650 (26.0) | 34190 (16.1) | 82720 (35.6) | 93750 (37.5) | 1754 (38.1) | 3136 (31.5)

12. Secondary Outcome: Observed Maximum Concentration (Cmax)
Description: To assess plasma pharmacokinetic parameters following single ascending doses of AZD977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Intellicap Device (Part B) | Oral Suspension (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 7 | 7
nmol/L | 201.6 (27.7) | 952.0 (20.9) | 3367 (41.3) | 5966 (40.6) | 7243 (27.7) | 7149 (17.2) | 14310 (29.1) | 16700 (29.2) | 161.2 (36.8) | 790.9 (22.9)

13. Secondary Outcome: Time to Maximum Observed Plasma Concentration (t Max)
Description: To assess plasma pharmacokinetic parameters following single ascending doses of AZD977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: as for outcome 10
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Intellicap Device (Part B) | Oral Suspension (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 7 | 7
Hour (h) | 0.50 [0.50 to 1.08] | 0.99 [0.50 to 1.02] | 0.50 [0.50 to 1.02] | 1.00 [0.48 to 1.00] | 0.88 [0.38 to 1.50] | 0.75 [0.50 to 1.00] | 3.51 [3.50 to 4.50] | 3.74 [2.50 to 4.50] | 4.02 [1.98 to 5.52] | 0.75 [0.23 to 1.50]

14. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t1/2λz)
Description: To assess plasma pharmacokinetic parameters following single ascending doses of AZD977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Intellicap Device (Part B) | Oral Suspension (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 2 | 5 | 4 | 4 | 7
Hour (h) | 1.741 (0.1753) | 1.755 (0.2923) | 7.161 (4.397) | 10.00 (1.933) | 9.618 (3.412) | 22.99 (6.527) | 21.17 (12.18) | 21.68 (3.495) | 11.60 (6.081) | 6.145 (3.365)

15. Secondary Outcome: Apparent Clearance (CL/F)
Description: To assess plasma pharmacokinetic parameters following single ascending doses of AZD977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Intellicap Device (Part B) | Oral Suspension (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 2 | 5 | 4 | 4 | 7
L/h | 24.52 (3.391) | 25.89 (5.546) | 28.46 (11.08) | 21.84 (5.812) | 28.49 (7.392) | 54.34 (19.16) | 20.99 (6.683) | 29.38 (8.430) | 45.97 (13.03) | 31.82 (10.79)

16. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: To assess plasma pharmacokinetic parameters following single ascending doses of AZD977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L
Groups:
- Part A - 400 mg AZD9977; Part A - 800 mg AZD9977: Subjects received 800 mg AZD9977, oral suspension under fasted conditions
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Intellicap Device (Part B) | Oral Suspension (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 2 | 5 | 4 | 4 | 7
L | 61.50 (9.724) | 64.52 (13.40) | 266.1 (180.6) | 315.8 (111.9) | 401.9 (180.0) | 1712 (123.7) | 652.5 (414.0) | 897.0 (210.6) | 720.1 (348.2) | 269.4 (142.2)

17. Secondary Outcome: Cumulative Amount of Unchanged Drug Excreted Into Urine [Ae (0-48)]
Description: To assess urine pharmacokinetic parameters following single ascending doses of AZD9977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 5
nmol | 2491 (213.4) | 12440 (2818) | 59700 (21910) | 122800 (27020) | 189700 (46420) | 178600 (32530) | 428600 (93430) | 503400 (132300)

18. Secondary Outcome: Fraction Excreted Unchanged in Urine[Fe (0-48)]
Description: To assess percentage of the total drug excreted in the urine that was unchanged following single ascending doses of AZD9977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 5
Percentage | 19.90 (1.705) | 19.88 (4.502) | 23.84 (8.750) | 24.53 (5.396) | 18.94 (4.635) | 8.917 (1.624) | 21.40 (4.664) | 16.75 (4.402)

19. Secondary Outcome: Renal Clearance of Drug From Plasma [CLR (0-48)]
Description: To assess urine pharmacokinetic parameters following single ascending doses of AZD9977
Time Frame: Pre-dose and post-dose upto 48 hrs
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 5
L/h | 5.018 (0.5818) | 5.061 (1.195) | 6.114 (1.533) | 5.230 (1.028) | 5.371 (0.6880) | 5.700 (1.097) | 5.274 (0.9817) | 5.319 (0.5086)

ADVERSE EVENTS:
Time Frame: SAEs will be collected from the signing of informed consent and AEs from randomization until the final follow-up visit in Part A, and from first dosing until the final follow-up visit in Part B.
Arm/Group | Part A- Placebo | Part A - 5 mg AZD9977 | Part A - 25 mg AZD9977 | Part A - 100 mg AZD9977 | Part A - 200 mg AZD9977 | Part A - 400 mg AZD9977 | Part A - 800 mg AZD9977 | Part A - 800 mg AZD9977 (Split Doses) | Part A - 1200 mg AZD9977 (Split Doses) | Part B
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/5 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 7/16 | 1/6 | 2/6 | 2/6 | 1/5 | 1/6 | 0/5 | 2/6 | 1/6 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A- Placebo (N=16) | Part A - 5 mg AZD9977 (N=6) | Part A - 25 mg AZD9977 (N=6) | Part A - 100 mg AZD9977 (N=6) | Part A - 200 mg AZD9977 (N=5) | Part A - 400 mg AZD9977 (N=6) | Part A - 800 mg AZD9977 (N=5) | Part A - 800 mg AZD9977 (Split Doses) (N=6) | Part A - 1200 mg AZD9977 (Split Doses) (N=6) | Part B (N=8)
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Backpain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.